CLINICAL TRIAL: NCT04268550
Title: A Phase II Study of LOXO-292 in Patients With RET Fusion-Positive Stage IV or Recurrent Non-Small Cell Lung Cancer (LUNG-MAP Sub-Study)
Brief Title: Targeted Treatment for RET Fusion-Positive Advanced Non-Small Cell Lung Cancer (A LUNG-MAP Treatment Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1900B; NCI-2019-08097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1900B (Other: SWOG); S1900B (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2020-01-08; First posted 2020-02-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selpercatinib) (Experimental): Patients receive selpercatinib orally PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Selpercatinib

INTERVENTIONS:
Drug: Selpercatinib — Given PO
  Other Names: LOXO-292; RET Kinase Inhibitor LOXO-292

SUMMARY:
This phase II LUNG-MAP treatment trial studies how well selpercatinib works in treating patients with RET fusion-positive non-small cell lung cancer that is stage IV or has come back (recurrent). Selpercatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the objective response rate (ORR) (confirmed complete or partial response) by blinded independent centralized review (BICR) associated with selpercatinib (LOXO-292) in patients with previously-treated stage IV or recurrent RET fusion-positive non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To evaluate the duration of BICR-assessed response among BICR responders. II. To evaluate the frequency and severity of toxicities. III. To evaluate the investigator-assessed objective response rate (confirmed complete or partial response).

IV. To evaluate duration of investigator-assessed response among patients with a response as determined by the local investigator.

V. To evaluate investigator-assessed progression-free survival (IA-PFS). VI. To evaluate BICR-assessed PFS. VII. To evaluate overall survival (OS).

VIII. Among patients with brain metastases at baseline:

VIIIa. To evaluate the central nervous system (CNS) response rate (confirmed complete response [CR]).

VIIIb. To evaluate the duration of intracranial response among patients with a CNS response.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To collect, process, and bank cell-free deoxyribonucleic acid (cfDNA) at baseline, progression, and end of treatment for future development of a proposal to evaluate comprehensive next-generation sequencing of circulating tumor deoxyribonucleic acid (ctDNA).

II. To establish a tissue/blood repository from patients with refractory non-small cell lung cancer (NSCLC).

OUTLINE:

Patients receive selpercatinib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years and then at the end of 3 years from date of sub-study registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been assigned to S1900B based on biomarker analysis of tissue and/or blood and determined to have RET fusion-positive NSCLC as defined here:

  * Patients must have RET fusion-positive NSCLC as determined by the Foundation Medicine (FMI) tissue-assay, other tumor-based assays such as next-generation sequencing (NGS), polymerase chain reaction (PCR), or follicular in situ hybridization (FISH), or by cfDNA blood assay. Patients with RET fusions detected by immunohistochemistry (IHC) alone are not eligible. The testing must be done within a laboratory with Clinical Laboratory Improvement Act (CLIA), International Organization for Standardization (ISO/International Electrotechnical Commission (IEC), College of American Pathologists (CAP), or similar certification. Presence of RET fusions detected on tests performed outside of LUNGMAP must have been confirmed by the study biomarker review panel
* For patients whose prior therapy was for stage IV or recurrent disease, the patient must have received at least one line of a platinum-based chemotherapy regimen. For patients whose prior systemic therapy was for stage I-III disease only (i.e. patient has not received any treatment for stage IV or recurrent disease), disease progression on platinum-based chemotherapy must have occurred within one year from the last date that the patient received that therapy. Prior anti-PD-1/PD-L1 therapy, alone or in combination (e.g. nivolumab, pembrolizumab, or durvalumab) is allowed
* Patients must be negative for all additional validated oncogenic drivers that could cause resistance to LOXO-292 treatment. This includes EGFR sensitizing mutations, EGFR T790M, ALK gene fusion, ROS1 gene fusion, KRAS activating mutation, BRAF V600E mutation and MET exon 14 skipping mutation or high-level amplification and expression

  * Note: EGFR, ALK, ROS, KRAS, and BRAF testing is performed as part of the LUNGMAP screening/pre-screening FoundationOne test. If prior data is not available, results from the FMI testing must be obtained prior to sub-study registration
* Patients must have measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI). The CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality. Measurable disease must be assessed within 28 days prior to sub-study registration. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 42 days prior to sub-study registration. All disease must be assessed and documented on the Baseline Tumor Assessment Form. Patients whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to registration. CT and MRI scans must be submitted for central review via transfer of images and data (TRIAD)
* Patients must have a CT or MRI scan of the brain to evaluate for CNS disease within 42 days prior to sub-study registration
* Patients with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on suppressive therapy within 28 days prior to registration
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. Patients with HCV infection who are currently on treatment must have an undetectable HCV viral load within 28 days prior to registration
* Patients with known human immunodeficiency virus (HIV) infection are eligible, provided they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 6 months prior to registration
* Patients must be able to swallow capsules
* Patients must have progressed (in the opinion of the treating physician) following the most recent line of therapy
* Patients must have recovered (=< grade 1) from any side effects of prior therapy. Patients must not have received any radiation therapy within 14 days prior to sub-study registration
* Absolute neutrophil count (ANC) >= 1,500/mcl (obtained within 28 days prior to sub-study registration)
* Platelet count >= 100,000 mcl (obtained within 28 days prior to sub-study registration)
* Serum bilirubin =< institutional upper limit of normal (IULN) (within 28 days prior to sub-study registration). For patients with liver metastases, bilirubin must be =< 5 x IULN
* Either alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 2 x IULN (within 28 days prior to sub-study registration) (if both ALT and AST are done, both must be =< 2 IULN). For patients with liver metastases, bilirubin and either ALT or AST must be =< 5 x IULN (if both ALT and AST are done, both must be =< 5 x IULN)
* Serum creatinine =< the IULN or calculated creatinine clearance >= 50 mL/min using the following Cockcroft-Gault formula (within 28 days prior to sub-study registration)
* Patients must have Zubrod performance status 0-1 documented within 28 days prior to sub-study registration
* Pre-study history and physical exam must be obtained within 28 days prior to sub-study registration
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Patients must have electrolytes and blood urea nitrogen (BUN) performed within 14 days prior to sub-study registration
* Patients must agree to have blood specimens submitted for circulating tumor DNA (ctDNA)
* Patients must also be offered participation in banking and in the correlative studies for collection and future use of specimens
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Patients with impaired decision-making capacity are eligible as long as their neurological or psychological condition does not preclude their safe participation in the study (e.g., tracking pill consumption and reporting adverse events to the investigator)

Exclusion Criteria:

* Patients must not have received any prior treatment with selective anti-RET inhibitors (anti-RET multikinase inhibitors are permitted)
* Patient must not have leptomeningeal disease, spinal cord compression or brain metastases unless: (1) metastases have been locally treated and have remained clinically controlled and asymptomatic for at least 14 days following treatment, and prior to registration, AND (2) patient has no residual neurological dysfunction and has been off corticosteroids for at least 24 hours prior to sub-study registration
* Patients must not have received any prior systemic therapy (systemic chemotherapy, immunotherapy or investigational drug) within 14 days prior to sub-study registration
* Patients must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment while receiving treatment on this study. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable
* Patient must not have had a major surgery within 14 days prior to sub-study registration. Patient must have fully recovered from the effects of prior surgery in the opinion of the treating investigator
* Patients must not have any grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., patients with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia
* Patients must not have a QT interval by Fridericia (QTcF) > 470 msec based on the electrocardiogram (ECG) within 28 days prior to registration. It is suggested that a local cardiologist review the QTcF intervals
* Patients must not have any clinically significant uncontrolled systemic illness, including but not limited to uncontrolled infection, requiring intravenous antibiotics, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmias, uncontrolled hypertension, or uncontrolled diabetes mellitus

  * Uncontrolled diabetes: Patients who have a diagnosis of diabetes must have an hemoglobin (Hb) A1C < 7% within 28 days prior to registration. The same criterion will be used in patients with confirmed diagnosis of diabetes mellitus who have been on a stable dietary or therapeutic regimen for this condition in the last three months
  * Uncontrolled blood pressure and hypertension: All blood pressure measurements within the 28 days prior to registration must be systolic blood pressure (SBP) =< 180 and diastolic blood pressure (DBP) =< 100. An exception can be made by a healthcare provider for a patient with a single blood pressure elevation who upon rechecking has a blood pressure within the parameters above
* Patients must not have any impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of LOXO-292 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or active peptic ulcer disease)
* Patients must not be planning to receive any strong inhibitors or inducers of CYP3A4 at least 14 days prior to sub-study registration and throughout protocol treatment
* Patients must not be planning to use proton pump inhibitors (PPIs) at least one week prior to sub-study registration and throughout protocol treatment
* Patients must not be pregnant or nursing. Women study patients of reproductive potential and fertile men study patients and their partners must abstain or use effective contraception (including barrier method) while receiving study treatment and for at least 3 months after the last dose of LOXO-292. Male study patients must agree not to donate sperm for 6 months after the last dose of LOXO-292. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Response rate by blinded independent centralized review (BICR) | Up to 3 years from date of sub-study registration
  A response will be confirmed by a complete response (CR) or partial response (PR). Proportions and associated confidence intervals will be calculated.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 3 years from date of sub-study registration
  Will be assessed using Common Terminology Criteria for Adverse Event version 5.0.
BICR-progression-free survival (PFS) | From date of sub-study registration to date of first documentation of progression assessed by BICR or symptomatic deterioration, or death due to any cause, assessed up to 3 years from date of sub-study registration
  Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to estimate confidence intervals for the median using Greenwood's formula and based on a log-log transformation applied on the survival function for landmark times
Investigator-assessed (IA) PFS | From date of sub-study registration to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause, assessed up to 3 years from date of sub-study registration
  Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to estimate confidence intervals for the median using Greenwood's formula and based on a log-log transformation applied on the survival function for landmark times
Overall survival | Up to 3 years from date of sub-study registration
  Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to estimate confidence intervals for the median using Greenwood's formula and based on a log-log transformation applied on the survival function for landmark times
BICR-duration of response (DOR) | From date of first documentation of confirmed response (CR or PR) to date of first documentation of progression assessed by BICR or symptomatic deterioration, or death due to any cause among patients who achieve, assessed at 6 and 12 months
  Will be evaluated among patients who achieve a confirmed response. Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to estimate confidence intervals for the median using Greenwood's formula and based on a log-log transformation applied on the survival function for landmark times. The median DOR and percentage with DOR at landmark times at 6 and 12 months after documentation of confirmed response will be estimated.
Central nervous system (CNS) response rate | Baseline
  Will be assessed among patients with brain metastases. Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to estimate confidence intervals for the median using Greenwood's formula and based on a log-log transformation applied on the survival function for landmark times
Duration of intracranial response among patients with a CNS response | Baseline
  Will be assessed among patients with brain metastases. Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to estimate confidence intervals for the median using Greenwood's formula and based on a log-log transformation applied on the survival function for landmark times

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Y Elamin, Principal Investigator — SWOG Cancer Research Network
Locations (306):
- United States (306):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Genesis Cancer Center - Silvis, Silvis, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Cancer Care Institute, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - HaysMed University of Kansas Health System, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Western Maryland Regional Medical Center, Cumberland, Maryland
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - University of Rochester, Rochester, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Rex Hematology Oncology Associates-Cary, Cary, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Rex Hematology Oncology Associates-Garner, Garner, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Rex Hematology Oncology Associates-Blue Ridge, Raleigh, North Carolina
  - Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Jefferson Healthcare, Port Townsend, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin